CLINICAL TRIAL: NCT01321164
Title: Fumaric Acid Esters Versus Fumaric Acid Esters Plus Narrow Band Type B Ultraviolet (UVB) in Patients With Severe Plaque Psoriasis
Brief Title: Fumaric Acid Versus Fumaric Acid Plus Narrow Band Type B Ultraviolet (UVB) for Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Adrian Tanew, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPUVB 005
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Fumarates; fumaric acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fumaric acid esters (Active Comparator): Fumaric acid esters monotherapy
  Interventions: Drug: Fumaric acid esters
- fumaric acid esters plus narrow band UVB (Experimental): Combination therapy of fumaric acid esters plus narrow band type B ultraviolet therapy (UVB)
  Interventions: Device: Full Body UV Therapy System UV 7002 plus fumaric acid esters

INTERVENTIONS:
Device: Full Body UV Therapy System UV 7002 plus fumaric acid esters — Combination therapy of narrow band type B ultraviolet (UVB) therapy plus fumaric acid esters therapy.
  Narrow band UVB therapy: 3 times a week for 6 weeks; Fumaric acid esters therapy: Capsules, schema therapy, 1 to 3 times a day for 6 months
  Other Names: TL-01;; Irradiation therapy with narrow band UVB
  Arms: fumaric acid esters plus narrow band UVB
Drug: Fumaric acid esters — Monotherapy, Capsules, schema therapy, 1 to 3 times a day, 6 months
  Other Names: Fumaric acid
  Arms: Fumaric acid esters

SUMMARY:
The main objective of the study is to evaluate the additional effect of a narrow band Type B Ultraviolet (UVB) therapy on the treatment of severe plaque psoriasis with fumaric acid esters (FAE) in comparison to FAE monotherapy. The secondary objectives are to evaluate the effect of an additional narrow band UVB therapy on the cumulative FAE dose required to reach Psoriasis Area and Severity Index (PASI) 75 in comparison to FAE monotherapy and to evaluate whether a leukopenia and lymphopenia frequently occurring during the FAE treatment is a positive predictive factor for the treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patient with moderately severe to severe Psoriasis (BSA ≥ 10 and PASI ≥ 10)
* Age between 18 and 80 years old

Exclusion Criteria:

* pregnant woman and satisfying women
* cancer, chronic infections, autoimmune diseases
* gastrointestinal illnesses
* liver diseases
* renal malfunctions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mean reduction in Psoriasis Area and Severity Index (PASI) | Baseline and 6 weeks

SECONDARY OUTCOMES:
Mean cumulative FAE dose required to reach PASI 75 | 6 months
Mean reduction in Psoriasis Area and Severity Index (PASI) | Baseline and 6 months
Mean reduction in Psoriasis Log-based Area and Severity Index (PLASI) | Baseline and 6 months
Mean reduction in Dermatology Life Quality INDEX (DLQI) | Baseline and 6 months
Mean white blood cells (Leukocytes and Lymphocytes) count | Baseline and 6 months
  Correlation between the mean white blood cells (Leukocytes and Lymphocytes) count and PASI reduction and between the mean white blood cells count and cumulative FAE dose.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Tanew, Prof. Dr., Principal Investigator — Medical University of Vienna, Department of Dermatology, Division of General Dermatology
Locations (1):
- Medical University of Vienna; Department of Dermatology, Vienna, Austria